CLINICAL TRIAL: NCT06897319
Title: Impact of High-Flow Tracheal Therapy on the Rheological Properties of Tracheobronchial Secretions in Tracheostomized Patients: A Randomized Crossover Study.
Brief Title: High-Flow Tracheal Therapy on Tracheobronchial Secretions in Tracheostomized Patients
Acronym: TRACH2O
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, William Poncin, PT, PhD, Principal Investigator, Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: TRACH2O
Record Dates: First submitted 2025-03-15; First posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Tracheostomized Patients

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFT (Experimental)
  Interventions: Device: High-Flow Tracheal Therapy
- Control (No Intervention)

INTERVENTIONS:
Device: High-Flow Tracheal Therapy — Device: Airvo 2 (Fisher & Paykel Healthcare) Settings: Flow rate start at 40L/min and will be adapted according to tolerance; temperature aimed at 37°C or 34°C according to tolerance, FiO₂ set (if needed) according to SpO2 target values.
  Arms: HFT

SUMMARY:
This monocentric, randomized crossover study aims to assess the impact of high-flow tracheal therapy (HFT) on the rheological properties of tracheobronchopulmonary secretions in tracheostomized patients. The primary objective is to compare the viscoelastic characteristics of secretions collected with and without HFT. Secondary objectives include evaluating the effects of HFT on dyspnea, patient comfort, and secretion appearance. The study will take place at Cliniques Universitaires Saint-Luc, with adult tracheostomized patients undergoing standard care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Tracheostomized patients
* Patients requiring routine tracheal suctioning and already using HFT overnight

Exclusion Criteria:

* Insufficient secretions for analysis
* Cognitive impairment or confusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-03-20 (Estimated); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Critical stress (σc) | Measured three times: at baseline, after one hour, after 4 hours
  The rheological properties measured using Rheomuco (Rheonova) will be sampled during a suctioning procedure.
  The critical stress σc = G*(γc).γc, where G*(γc) is the viscoelastic modulus measured at the critical strain, is the measured stress at which this transition occurs.
  See the description of the other rheological outcomes in the secondary outcomes.

SECONDARY OUTCOMES:
Dyspnea (modified Borg scale) | Measured two times: at baseline and after 4 hours
  The modified Borg Scale (from 0 : no dyspnea; to 10 : maximal dyspnea) will be used
Patient Comfort (Visual Analog Scale - VAS) | Measured two times: at baseline and after 4 hours
  The VAS (from 0 : extremely comfortable; to 10 : extremely uncomfortable) will be used
Secretion Appearance (Murray Scale) | Measured two times: at baseline and after 4 hours
  The Murray scale define the following secretion appearance:
  * Mucoid
  * Mucopurulent
  * Purulent
Viscoelastic modulus (G*) | Measured three times: at baseline, after one hour, after 4 hours
  The rheological properties measured using Rheomuco (Rheonova) will be sampled during a suctioning procedure.
  The ratio of the stress to the strain, the viscoelastic modulus G* , describes the molecular network force in response to shear.
  In viscoelastic materials, the viscous dissipation shifts in time the stress response to the imposed strain, which is quantified by the damping ratio tan δ. Both G* and tan δ provide the viscous and elastic moduli, G' and G''.
  See the description of the other rheological outcomes in the secondary outcomes.
Damping ratio (tan δ) | Measured three times: at baseline, after one hour, after 4 hours
  The rheological properties measured using Rheomuco (Rheonova) will be sampled during a suctioning procedure.
  At given deformation, a damping ratio above 1 would describe a predominantly viscous material (G'' > G'), i.e. that behaves like a liquid, whereas a damping ratio below 1 denotes a predominantly elastic material (G' > G''), that exhibits a solid-like behavior.
Critical strain (γc) | Measured three times: at baseline, after one hour, after 4 hours
  The rheological properties measured using Rheomuco (Rheonova) will be sampled during a suctioning procedure.
  The viscoelastic characteristics are measured at increasing strains, ranging from about 1 % to about 10000 %. At a critical strain value, γc, typically around or above 1000 % for sputa, the G' and G'' curves cross over (the damping ratio overcomes 1). Beyond this critical point, the sample becomes predominantly viscous over elastic (fluid-like) under strain and starts to flow.
  See the description of the other rheological outcomes in the secondary outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques universitaires Saint-Luc, Brussels, Belgium